CLINICAL TRIAL: NCT03762252
Title: Effects of Dry Needling of Active Trigger Points in the Scalene Muscles on Individuals With Mechanical Neck Pain
Brief Title: Dry Needling of Scalene Muscle Trigger Points in Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Director of Department, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC 2018-12-10
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Patients will receive dry needling over active trigger points in the scalene muscles
  Interventions: Other: Dry needling
- Manual Therapy (Active Comparator): Patients will receive a manual compression for 30seconds over active trigger points in the scalene muscles
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Dry needling — A solid filiform needle will be inserted over active trigger points in the scalene muscles for 30 seconds. The aim will be to elicit local twitch responses or the referred pain pattern of the scalene muscles.
  Arms: Dry needling
Other: Manual Therapy — The therapist will apply manual compression over active trigger points in the scalene muscles for 30 seconds
  Arms: Manual Therapy

SUMMARY:
There is preliminary evidence suggesting that referred pain from active trigger points can play a relevant role in individuals with mechanical neck pain. Some studies have investigated the effectiveness of dry needling over the upper trapezius muscle in this population. However, other muscles, such as the scalene muscles, can be also relevant for neck pain symptoms. No study has investigated the effects of the application of dry needling over active trigger points in the scalenes muscles in a sample of patients with mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

Generalized neck-shoulder pain with symptoms provoked by neck postures, neck movement, or palpation of the cervical musculature

Exclusion Criteria:

* whiplash injury;
* previous cervical or thoracic surgery;
* cervical radiculopathy or myelopathy;
* diagnosis of fibromyalgia syndrome;
* having undergone physical therapy in the previous 6 months;
* less than 18 or greater than 45 years of age
* fear to needles
* any respiratory disease, e.g., chronic brochitis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in neck pain intensity with a numerical pain rate scale before and after the intervention | Baseline, one day (immediately post), 7 days (one week) and 30 days (one month) after the intervention
  A Numerical Pain Rate Scale (NPRS, 0-10) will be used to assess spontaneous neck pain intensity

SECONDARY OUTCOMES:
Changes in oxigen saturation with a pulse oximeter before and after the intervention | Baseline, one day (immediately post), 7 days (one week) and 30 days (one month) after the intervention
  Oxygen saturation will be monitored with a handheld pulse oximeter with Masimo SET® measure-through Motion and Low Perfusion™ pulse oximeter
Changes in inspiratory vital capacity with an incentive spirometer before and after the intervention | Baseline, one day (immediately post), 7 days (one week) and 30 days (one month) after the intervention
  Changes in inspiratory vital capacity will be assessed with the incentive spirometer DHD Coach 2®
Changes in neck-related disability with the Neck Disability Index before and after the intervention | Baseline and 7 days (one week) and 30 days (one month) after the intervention
  The Neck Disability Index (NDI, 0-50), a specific neck pain related disability questionaire, will be used for assessing neck pain related-disability

CONTACTS AND LOCATIONS:
Overall Officials: César Fernández-de-las-Peñas, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- César Fernández-de-las-Peñas, Alcorcón, Madrid, Spain